CLINICAL TRIAL: NCT00005467
Title: Indices of Severity and Prognosis for Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4912; R01HL042498 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Anemia, Sickle Cell; Blood Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases

SUMMARY:
To develop a clinical severity index that could prospectively identify sickle cell disease patients who were at high risk for a turbulent clinical course and a poor prognosis.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Using the database, univariate analysis showed that factors associated with the occurrence of cerebrovascular accident (51 patients) included hematocrit, rate of change of pocked red cell count, and polymer fraction at 40 percent oxygen saturation (PF40). Only low hematocrit was predictive of death in the pediatric cohort. There were 45 disease-related deaths.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-01; Study Completion 1992-12 (Actual)

REFERENCES:
- [Background] Bray GL, Muenz L, Makris N, Lessin LS. Assessing clinical severity in children with sickle cell disease. Preliminary results from a cooperative study. Am J Pediatr Hematol Oncol. 1994 Feb;16(1):50-4. PMID 8311173